CLINICAL TRIAL: NCT01256411
Title: An Open-label, Long-term Extension Study to Evaluate the Safety, Tolerability and Efficacy of 12 Months of LCZ696 Treatment in Patients With Essential Hypertension
Brief Title: A Long-term (12 Months) Safety, Tolerability and Efficacy Study of LCZ696 in Patients With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCZ696A2219E1
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Essential Hypertension
Keywords: hypertension; blood pressure; LCZ696; dual-acting; neprilysin; nep inhibitor; vasopeptidase; angiotensin receptor; angiotensin receptor neprilysin inhibitor (ARNi)
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; Amlodipine; Hydrochlorothiazide

ARMS (1):
- LCZ696 (Experimental)
  Interventions: Drug: LCZ696; Drug: Amlodipine; Drug: Hydrochlorothiazide (HCTZ)

INTERVENTIONS:
Drug: LCZ696 — Participants received LCZ696 200 mg as the starting dose with optional down titration to 100 mg for tolerance and optional up titration to 400 mg for adequate blood pressure control.
Drug: Amlodipine — Optional add-on of amlodipine (5-10 mg) was allowed (as applicable per local country regulations) for adequate blood pressure control.
Drug: Hydrochlorothiazide (HCTZ) — Optional add-on of hydrochlorothiazide (HCTZ) (12.5-25 mg) was allowed (as applicable per local country regulations) for adequate blood pressure control.

SUMMARY:
The purpose of this study is to assess the long-term safety, tolerability and efficacy of LCZ696.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have successfully completed protocol No. CLCZ696A2219 and who, as judged by the study investigator, are able to continue in the current study.
* Ability to communicate and comply with all study requirements and demonstrate good medication compliance during CLCZ696A2219.

Exclusion Criteria:

* Patients who did not complete CLCZ696A2219.
* Presence of significant protocol violation in CLCZ696A2219.
* Patients who are deemed to be unable to comply with the protocol by the investigator.
* Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- China (5):
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Tianjin
- Japan (10):
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Kunitachi, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- South Korea (5):
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Koyang, Kyunggi
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Seoul
- Taiwan (3):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Changhua
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Analyses on this open label extension study were performed according to treatment groups defined by the maximum and highest dose treatments received: 1) LCZ696 200 mg, 2) LCZ696 400 mg, 3) LCZ696 400 mg/Amlodipine, 4) LCZ696 400 mg/Amlodipine/HCTZ, 5) LCZ696 Mono (LCZ696 only), and 6) LCZ696 Combination LCZ696 with Amlodipine and/or HCTZ).
Groups:
- LCZ696 200 mg: Participants received LCZ696 200 mg by mouth once daily (qd).
- LCZ696 400 mg: Participants received LCZ696 400 mg by mouth qd.
- LCZ606 400 mg/Amlodipine: Participants received LCZ696 400 mg by mouth qd and amlodipine 5mg up to 10 mg by mouth as needed (prn).
- LCZ696 400 mg/Amlodipine/HCTZ: Participants received LCZ696 400 mg by mouth qd, amlodipine 5 mg up to 10 mg by mouth prn and HCTZ 6.25 mg and up to 25 mg by mouth prn.
- LCZ696 Monotherapy: Participants received LCZ696 only.
- LCZ696 Combination Therapy: Participants received LCZ696 with amlodipine and/or HCTZ.
Period: Extension by Maximum Treatment
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ606 400 mg/Amlodipine | LCZ696 400 mg/Amlodipine/HCTZ | LCZ696 Monotherapy | LCZ696 Combination Therapy
Started | 139 | 89 | 109 | 4 | 0 | 0
Down Titrated to 100 mg | 12 | 0 | 0 | 0 | 0 | 0
Completed | 132 | 79 | 105 | 4 | 0 | 0
Not Completed | 7 | 10 | 4 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 6 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 2 | 1 | 0 | 0 | 0
Period: Extension by Mono or Combination Therapy
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ606 400 mg/Amlodipine | LCZ696 400 mg/Amlodipine/HCTZ | LCZ696 Monotherapy | LCZ696 Combination Therapy
Started | 0 | 0 | 0 | 0 | 228 | 113
Completed | 0 | 0 | 0 | 0 | 211 | 109
Not Completed | 0 | 0 | 0 | 0 | 17 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 6 | 1
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 7 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ606 400 mg/Amlodipine | LCZ696 400 mg/Amlodipine/HCTZ | Total
Number analyzed (Participants) | 139 | 89 | 109 | 4 | 341
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (9.69) | 50.3 (10.14) | 52.5 (9.53) | 46.3 (2.06) | 51.8 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 18 | 26 | 0 | 99
  Male | 84 | 71 | 83 | 4 | 242

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, and Deaths (Analysis by Actual Treatment)
Description: Participants were monitored throughout the study for adverse events, serious adverse events and deaths.
Time Frame: Baseline to 12 months
Population: Actual extension treatment received: The participants are included in each treatment group for which they received treatment. For example, if a participant started on LCZ696 200 mg but was then down-titrated to LCZ696 100 mg, the participant was counted once in the LCZ696 100 mg group and once in the LCZ696 200 mg group.
Measure: Number; unit: Participants
Groups:
- LCZ696 100 mg: Participants were down-titrated to 100 mg.
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ606 400 mg/Amlodipine | LCZ696 400 mg/Amlodipine/HCTZ | LCZ696 100 mg
Number analyzed (Participants) | 340 | 201 | 112 | 4 | 12
Participants
  Adverse events (serious and non-serious) | 147 | 78 | 53 | 0 | 6
  Seroius adverse events | 10 | 2 | 0 | 0 | 1
  Deaths | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) and Mean Sitting Diastolic Blood Pressure (msDBP) (Analysis by Maximum Treatment)
Description: Sitting BP measurements were performed at every study visit. A negative change from baseline indicates improvement.
Time Frame: Baseline, 12 months
Population: Treated set: The treated set included all participants who received at least one dose of extension study medication. One participant in the LCZ696 400 mg/Amlodopine group discontinued after 1 day in the extension study without having any BP measurements taken during the extension. Therefore, this participant was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ606 400 mg/Amlodipine | LCZ696 400 mg/Amlodipine/HCTZ
Number analyzed (Participants) | 139 | 89 | 108 | 4
mmHg
  msDBP | -16.6 (7.63) | -14.2 (7.05) | -17.4 (7.71) | -16.8 (3.84)
  msSBP | -24.1 (12.16) | -21.3 (11.46) | -28.1 (13.43) | -29.0 (9.23)

3. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) and Mean Sitting Diastolic Blood Pressure (msDBP) (Analysis by Mono or Combination Therapy)
Description: Sitting BP measurements were performed at every study visit. A negative change from baseline indicates improvement.
Time Frame: Baseline, 12 months
Population: Treated set: The treated set included all participants who received at least one dose of extension study medication. One participant in the LCZ696 combination group discontinued after 1 day in the extension study without having any BP measurements taken during the extension. Therefore, this participant was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 Monotherapy | LCZ696 Combination Therapy
Number analyzed (Participants) | 228 | 112
mmHg
  msDBP | -15.7 (7.49) | -17.3 (7.60)
  msSBP | -23.0 (11.95) | -28.2 (13.27)

4. Secondary Outcome: Number of Participants With Blood Pressure Control Rate of <140/90 mmHg (Analysis by Maximum Treatment)
Description: Blood pressure (BP) control is defined as BP <140/90 mmHg.
Time Frame: Baseline to 12 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | LCZ606 400 mg/Amlodipine | LCZ696 400 mg/Amlodipine/HCTZ
Number analyzed (Participants) | 139 | 89 | 108 | 4
Participants | 114 | 62 | 77 | 3

5. Secondary Outcome: Number of Participants With Blood Pressure Control Rate of <140/90 mmHg (Analysis by Mono or Combination Therapy)
Description: Blood pressure (BP) control is defined as BP <140/90 mmHg.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | LCZ696 Monotherapy | LCZ696 Combination Therapy
Number analyzed (Participants) | 228 | 112
Participants | 176 | 80

ADVERSE EVENTS:
Groups:
- LCZ696 400 mg/Aml; LCZ696 400 mg/Aml/HCTZ: Participants received LCZ696 400 mg by mouth qd, amlodipine 5 mg up to 10 mg by mouth prn and HCTZ 6.25 mg and up to 25 mg by mouth prn.
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | LCZ696 400 mg/Aml | LCZ696 400 mg/Aml/HCTZ
Serious Adverse Events (participants affected / at risk) | 1/12 | 10/340 | 2/201 | 0/112 | 0/4
Other Adverse Events (participants affected / at risk) | 6/12 | 77/340 | 39/201 | 32/112 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 100 mg (N=12) | LCZ696 200 mg (N=340) | LCZ696 400 mg (N=201) | LCZ696 400 mg/Aml (N=112) | LCZ696 400 mg/Aml/HCTZ (N=4)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 100 mg (N=12) | LCZ696 200 mg (N=340) | LCZ696 400 mg (N=201) | LCZ696 400 mg/Aml (N=112) | LCZ696 400 mg/Aml/HCTZ (N=4)
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Radicular cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 37 | 15 | 15 | 0
Pharyngitis (Infections and infestations) | 0 | 3 | 2 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 20 | 4 | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 5 | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 13 | 6 | 9 | 0
Headache (Nervous system disorders) | 2 | 6 | 2 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 5 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 3 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.